CLINICAL TRIAL: NCT03817255
Title: Identification of Excessive Substance Use to Encourage Behaviour Change Among Young People in Primary Care: Pilot Study in Preparation for a Randomized Trial
Brief Title: Young People's Health Assessment as Treatment and Health Guide
Acronym: YP-HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Prof. Dagmar M. Haller, Professor, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YP-HEALTH Pilot
Record Dates: First submitted 2019-01-08; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Adolescent Behavior; Substance Use
MeSH Terms: conditions — Adolescent Behavior; Substance-Related Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the intervention or the control condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants: Although they cannot be masked to the content of the intervention (questionnaire), they are only informed that the study is about health behaviours in general. Thus, they are masked as to whether they are in the intervention or control group.
  Care provider: As they cannot have access to the participants' questionnaires, they are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Substance use (Experimental): In this screening intervention, participants complete a substance use questionnaire (=intervention).
  Interventions: Other: Substance use questionnaire
- Physical activity (Active Comparator): In this screening control condition, participants complete a physical activity questionnaire (=control).
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Substance use questionnaire — Questions about substance use based on the Detection of Alcohol and Drug Problems in Adolescents (DEP-ADO) survey.
  Arms: Substance use
Other: Physical activity — Questions about physical activity, based on the short version of the International Physical Activity Questionnaire (IPAQ).
  Arms: Physical activity

SUMMARY:
Background: Excessive alcohol and other substance use in adolescence is prevalent and has developmental consequences that extend into adulthood. In parallel with other public health and clinical measures, early identification in primary care represents an important step to address this problem. Screening and brief intervention by primary care physicians is recommended but often fails to be implemented due to time constraints and other barriers. Working hypothesis: Recent evidence suggests that simply asking individuals about their substance use may in itself encourage behaviour change, regardless of the clinical intervention that may follow. This hypothesis has not as yet been tested in a population of young people consulting in primary care. The investigators hypothesise that inviting young people to complete a brief substance use screening questionnaire in the waiting room before their primary care consultation has the potential to lead to a decrease in substance use in the months following this consultation.

Specific aims: The aim of this pilot project is to develop and test the methods for a future randomized trial. The future trial will assess the effectiveness of pre-consultation substance use screening, compared to screening for other behaviors, on subsequent substance use in young people between the ages of 15 and 24 years consulting primary care physicians.

Expected value of the proposed project: The clinical context of primary care has the potential to trigger behavior change in young people, thus favoring improved adult outcomes in this population. If effective, pre-consultation substance use screening could contribute to a reduction in excessive substance use among young people in a simple and cost-effective way. This pilot study will provide precious feasibility data for the design of the related cluster randomised trial.

DETAILED DESCRIPTION:
Background:

Excessive alcohol and other substance use in adolescence has short and long term consequences on health and contributes extensively to lifelong morbidity. Since prevalence of this excessive use is high among young people consulting in primary care, primary care physicians (PCPs) are well placed to address this problem. PCPs are encouraged to screen and provide brief interventions addressing excessive substance use in young people, but a range of barriers, such as time constraints and insufficient training, limits the implementation of these recommendations in primary care practices. Several recent trials of brief primary care interventions showed substantial reductions in the proportion of participants who were excessive substance users at follow-up (20% to 30% reductions), but no statistically significant differences between the intervention and control groups. Reductions in substance use in the control group can be due to several factors: 1) Regression to the mean (repeat participant responses show a trend towards the mean values for the participating population), 2) Research participation effects (e.g. Hawthorne effect, social desirability bias), 3) Historical trends which affect the entire population, such as reductions in per capita alcohol use in relation to public health measures, 4) Assessment reactivity, when pre-intervention assessment itself encourages behavior change and thus serves as an intervention. In a randomized design these factors should apply equally to both groups, and additional effects of the tested intervention may still be visible. If reductions in substance use at follow-up are due to assessment reactivity, this suggests screening in the clinical context could act as an intervention in itself and be as effective as a brief intervention within the consultation. To date this hypothesis has not been explored in a population of young people attending primary care.

Aim of the Trial:

To assess the effectiveness of simply screening participants for excessive substance use before the consultation in the waiting room in reducing the prevalence of excessive substance use in young people attending primary care.

Objectives of the pilot study:

1. To pilot all methods for a randomized trial of the substance use screening intervention (patient recruitment, intervention and control conditions, follow-up procedures),
2. To obtain feedback from PCPs and patients in relation to the feasibility and acceptability of the proposed methods for the trial.

Methods:

The intervention screening questionnaire will be based on an instrument developed for previous trials. Questions for the control condition (about physical activity) will be based on a validated physical activity questionnaire (International Physical Activity Questionnaire, IPAQ). As recommended in guidelines for adolescent health and primary care research, both young people and PCPs will be involved in the development of the screening tools. A reference group of young people and of PCPs will be established in order to benefit from their input into the design of the study.

The intended trial procedure including recruitment of young people, screening for health risk behaviours and follow-up will be piloted in 6 primary care practices in the canton of Geneva in order to inform the final design of the trial.

The physicians involved in the advisory-group will be invited to undertake the pilot study in their own practices. They will be asked to include a minimum of five patients each. Patients will be randomized to either the intervention or the control questionnaire.

Patients will be recruited using a similar procedure as the one developed for one of our previous studies, the PRISM-Ado trial. Prior to the consultation, eligible patients will be invited by the practice assistant to participate in the study. Participants will be given an information and consent form, and will be given the choice to complete the study questionnaire either online (using a QR code to access the questionnaire on their phone) or in a paper format, in the waiting room. Participants will be asked to provide a contact phone number (mobile phone) to allow follow-up assessments 1 month following the consultation. Young people involved in the PRISM-Ado study underlined that they would be less likely to respond honestly to a screening questionnaire if it were to be used by the doctor in the consultation. Therefore this pre-consultation questionnaire will be entirely anonymous and will not be available for the PCPs to help them identify at-risk consumers. Written informed consent will be obtained from all young people before they complete the screening survey. Patient questionnaires will be coded to ensure anonymity.

A meeting of participating doctors will be organized to receive feed-back on all aspects of the study. Participating patients will be asked to provide their contact details (mobile phone number) so that they may be contacted to provide feed-back on the screening questionnaire and study procedure.

Physicians' and young people's characteristics will be summarized using frequencies for categorical data and means and standard deviations for continuous data. This summary will provide us with an initial profile of youth consulting in the practices and will inform planning and sample size calculations for the randomized trial. Participant feed-back will be summarized in a qualitative way.

Importance of the expected results:

The results of this pilot study will provide precious information for the final design of the randomised trial in primary care. These results will be published in a medical journal and presented at medical conferences. The consequences of excessive substance use in adolescence extend into adulthood. The investigators are hopeful that the interventions developed and piloted in this project will provide new ways of ensuring better health for young people today and in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting at the participating primary care practice during the recruitment period (2 months).

Exclusion Criteria:

* Acute illness requiring immediate attention of the physician
* Severe mental health conditions requiring treatment in a specialized setting
* Inability to read the trial information in French
* Person not consulting as a patient (e.g. parent of a child consulting a pediatrician, accompanying friend or partner).

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
The number of patients recruited by each PCP within a 2-month period | 2 months
  A maximum of 10 patients were to be recruited by each of the 6 participating primary care physicians (PCPs) within a 2-month period. The target number was 5 patients per PCP, but the recruitment period was not prolonged if this target was not met.
The proportion of PCPs who recruited at least 5 patients within a 2-month period | 2 months
  The participating PCPs were asked to recruit a minimum of 5 patients, but the recruitment period was limited to 2 months (for practical and financial reasons). All participating PCPs participated in the pilot study thinking that they would be able to recruit 5 patients. This outcome thus gives us an idea about whether PCPs had a realistic idea about their ability to recruit a sufficient number of eligible patients.
The proportion of eligible patients who agreed to participate | 2 months
  Measurement tool : A form completed by the PCPs assistants, documenting how many patients were approached, how many refused, and how many had exclusion criteria.
The proportion of PCPs who respected the pre-determined sequence of questionnaires (randomized sequence). | 2 months
  Each PCP received a unique randomized sequence of intervention and control questionnaires, in envelopes numbered from 1 to 10. At the end of the two-month recruitment period, they returned all envelopes (completed and empty questionnaires). The research team checked whether the sequence from 1 to 10 had been respected.
The proportion of participating patients who returned a completed baseline questionnaire (=patients included in study). | 2 months
  The PCPs did not check whether the questionnaires had been completed correctly (for confidentiality reasons). This proportion was thus determined by the research team. A questionnaire was considered "complete" if: 1. Consent form was signed, 2. Phone number was given, and 3. at least 50% of questions had been answered.
The proportion of patients included in the study who answered the follow-up questionnaire at one month. | 2 months
  Patients who could be contacted by phone one month after the baseline questionnaire, and who agreed to answer the second questionnaire (over the phone, with a member of the research team).
The proportion of patients at follow-up who consumed alcohol at least once in the last 30 days. | 2 months
  Patient self-report on follow-up telephone questionnaire. This outcome serves to ascertain that the study target group (= young people consuming alcohol or cannabis) can be reached through the study procedures.
The proportion of patients at follow-up who consumed cannabis at least once in the last 30 days. | 2 months
  Patient self-report on follow-up telephone questionnaire. This outcome serves to ascertain that the study target group (= young people consuming alcohol or cannabis) can be reached through the study procedures.

SECONDARY OUTCOMES:
The proportion of participants choosing to complete the paper questionnaire vs the online version. | 2 months
  Questionnaires were distributed in paper form, but could be filled in on a mobile device using a link (QR code).
Proportion of patients at follow-up stating that the procedures in the PC practices respected confidentiality. | 2 months
  At the end of the phone questionnaire, the researcher asked: " Did you feel that the procedures used in the study were confidential ? ", followed by an open question asking to elaborate on the context in which the questionnaire was completed (waiting room, presence of other patients/people).
PCPs critical comments regarding patient recruitment in their practices. | 1 month
  Narrative synthesis of meeting notes, collected during a group meeting with participating PCPs, by asking open-ended questions and open group discussion. PCPs were asked to describe difficulties with recruitment and to elaborate how these difficulties could be overcome, stimulating discussion and exchange within the group.

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar M Haller, Prof, Principal Investigator — University of Geneva
Locations (1):
- Primary Care Unit, University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available for this feasibility study for data protection reasons, because there will be a very limited number of participants.

REFERENCES:
- [Background] Haller DM, Meynard A, Lefebvre D, Hasselgard-Rowe J, Broers B, Narring F. Excessive substance use among young people consulting family doctors: a cross-sectional study. Fam Pract. 2015 Oct;32(5):500-4. doi: 10.1093/fampra/cmv058. Epub 2015 Aug 5. PMID 26251025
- [Background] Haller DM, Meynard A, Lefebvre D, Ukoumunne OC, Narring F, Broers B. Effectiveness of training family physicians to deliver a brief intervention to address excessive substance use among young patients: a cluster randomized controlled trial. CMAJ. 2014 May 13;186(8):E263-72. doi: 10.1503/cmaj.131301. Epub 2014 Mar 10. PMID 24616136
- [Background] Heather N. Interpreting null findings from trials of alcohol brief interventions. Front Psychiatry. 2014 Jul 16;5:85. doi: 10.3389/fpsyt.2014.00085. eCollection 2014. PMID 25076917
- [Background] McCambridge J, Kypri K. Can simply answering research questions change behaviour? Systematic review and meta analyses of brief alcohol intervention trials. PLoS One. 2011;6(10):e23748. doi: 10.1371/journal.pone.0023748. Epub 2011 Oct 5. PMID 21998626
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Haller DM, Meynard A, Lefebvre D, Tylee A, Narring F, Broers B. Brief intervention addressing excessive cannabis use in young people consulting their GP: a pilot study. Br J Gen Pract. 2009 Mar;59(560):166-72. doi: 10.3399/bjgp09X419529. PMID 19275832
- [Background] Sanci LA, Sawyer SM, Kang MS, Haller DM, Patton GC. Confidential health care for adolescents: reconciling clinical evidence with family values. Med J Aust. 2005 Oct 17;183(8):410-4. doi: 10.5694/j.1326-5377.2005.tb07104.x. PMID 16225445
- [Background] Haller DM, Sanci LA, Patton GC, Sawyer SM. Practical evidence in favour of mature-minor consent in primary care research. Med J Aust. 2005 Oct 17;183(8):439. doi: 10.5694/j.1326-5377.2005.tb07114.x. No abstract available. PMID 16225455